CLINICAL TRIAL: NCT05642091
Title: Role of Ultrasound Elastography in Pleural Effusion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mai Assem Abd-elkareem Aly, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Ultrasound Elastography
Record Dates: First submitted 2022-07-30; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transudate effusion (Active Comparator)
  Interventions: Device: ultrasound Elastography
- exudative effusion (Active Comparator)
  Interventions: Device: ultrasound Elastography

INTERVENTIONS:
Device: ultrasound Elastography — application of shear wave force by ultrasound elastography

SUMMARY:
Diagnostic performance of u.s elastography in pleural effusion

DETAILED DESCRIPTION:
Pleural fluid is an extremely common problem however the diagnosis of pleural effusion remain challenging due its diverse aetiologies .transthoracic ultrasound is often the initial tool to help diagnosis of pleural effusion.

Ultrasound elastography is a novel ultrasound technology that can differentiate malignant disease from benign disease by quantitatively assses tissue stifness by measuring the degree of distortion under application of an external force (shear wave ) However, very limited studies are available evaluating the efficacy of this novel technique in diagnosis of malignant pleural effusion.

ELIGIBILITY:
Inclusion Criteria:

.patients with pleural effusion above18 year

Exclusion Criteria:

* patients who refuse to undergone further investigations to reach final diagnosis of cause of pleural effusion

.patients with intercostal tube inserted in the effusion before enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-13 (Estimated); Primary Completion 2025-08-13 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
detect diagnostic performance of ultrasound elastography in pleural effusion | 3 months
  differentiate between elastisty index in benign and malignant pleural effuison that expressed in kpa by measuring it using ultrasound elastography

CONTACTS AND LOCATIONS:
Overall Officials: doaa mohamed magdy, associate prof, Study Director — assuit university hospital; sahar refaat mahmoud, lecturer, Study Director — assuit university hospital

REFERENCES:
- [Background] Hooper C, Lee YC, Maskell N; BTS Pleural Guideline Group. Investigation of a unilateral pleural effusion in adults: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii4-17. doi: 10.1136/thx.2010.136978. No abstract available. PMID 20696692
- [Background] Jiang B, Li XL, Yin Y, Zhang Q, Zang T, Song WS, Wang XM, Kang J, Herth FJF, Hou G. Ultrasound elastography: a novel tool for the differential diagnosis of pleural effusion. Eur Respir J. 2019 Aug 22;54(2):1802018. doi: 10.1183/13993003.02018-2018. Print 2019 Aug. PMID 31151959
- [Background] Davies CW, Gleeson FV, Davies RJ; Pleural Diseases Group, Standards of Care Committee, British Thoracic Society. BTS guidelines for the management of pleural infection. Thorax. 2003 May;58 Suppl 2(Suppl 2):ii18-28. doi: 10.1136/thorax.58.suppl_2.ii18. No abstract available. PMID 12728147
- [Background] Light RW, Macgregor MI, Luchsinger PC, Ball WC Jr. Pleural effusions: the diagnostic separation of transudates and exudates. Ann Intern Med. 1972 Oct;77(4):507-13. doi: 10.7326/0003-4819-77-4-507. No abstract available. PMID 4642731
- [Background] Bibby AC, Dorn P, Psallidas I, Porcel JM, Janssen J, Froudarakis M, Subotic D, Astoul P, Licht P, Schmid R, Scherpereel A, Rahman NM, Cardillo G, Maskell NA. ERS/EACTS statement on the management of malignant pleural effusions. Eur Respir J. 2018 Jul 27;52(1):1800349. doi: 10.1183/13993003.00349-2018. Print 2018 Jul. PMID 30054348
- [Background] Havelock T, Teoh R, Laws D, Gleeson F; BTS Pleural Disease Guideline Group. Pleural procedures and thoracic ultrasound: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii61-76. doi: 10.1136/thx.2010.137026. No abstract available. PMID 20696688